CLINICAL TRIAL: NCT04843982
Title: Effects of Esketamine Combined With Propofol for Sedation on Systemic Inflammation and Immune Function in Septic Patients in the ICU: a Single-center, Non-blind, Prospective Randomized Controlled Trial
Brief Title: Immunoinflammatory Regulation of Esketamine in Septic Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YSY202001
Record Dates: First submitted 2021-03-29; First posted 2021-04-14 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Esketamine; Sepsis; Inflammatory Response; Immunosuppression
Keywords: Esketamine; Sepsis; Inflammatory Response; Immunosuppression
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- esketamine plus propofol (Experimental): After inclusion, patients are sedated primarily with propofol (0-3 mg/kg/h) using a microinfusion pump and adjusted according to the depth of sedation (Richmond Agitation Sedation Scale (RASS): 0 to -2).
  After inclusion, septic patients will be received a single intravenous injection of esketamine (0.7 mg/kg), and then followed by an intravenous administration of esketamine (0.07 mg/kg/h) with an infusion pump for three consecutive days.
  Interventions: Drug: Esketamine hydrochloride
- propofol (No Intervention): After inclusion, patients are sedated primarily with propofol (0-3 mg/kg/h) using a microinfusion pump and adjusted according to the depth of sedation (Richmond Agitation Sedation Scale (RASS): 0 to -2).

INTERVENTIONS:
Drug: Esketamine hydrochloride — After inclusion, septic patients will be received a single intravenous injection of esketamine (0.7 mg/kg), and then followed by an intravenous administration of esketamine (0.07 mg/kg/h) with an infusion pump for three consecutive days.
  Arms: esketamine plus propofol

SUMMARY:
Studies have shown that excessive systemic inflammatory response and concomitant immunosuppression are the main cause of early death in patients with sepsis. Therefore, it is very important to reduce excessive inflammation and improve immunosuppression in the acute phase of sepsis. Clinical studies have shown that esketamine combined with propofol for sedation has been proven to be safe and effective for septic patients in the ICU due to its cardiovascular stability. Previous studies have demonstrated that esketamine has anti-inflammatory effects against depression and surgical stress. Our preliminary experimental studies have found that esketamine had strong anti-inflammatory effects in the acute phase of sepsis. However, it is not clear whether esketamine could reduce excessive inflammation and improve immunosuppression in septic patients primarily sedated with a continuous infusion of propofol.

This intervention study is to investigate whether three consecutive days of intravenous esketamine infusions via infusion pump (0.07 mg/kg/h) could reduce excessive inflammation and improve immunosuppression in septic patients requiring mechanical ventilation in the ICU under sedation primarily with propofol.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ age ≤60 years old;
* SOFA score ≥2;
* Mechanical ventilation should be required for at least 24 hours when included in the study;
* Informed consent is obtained.

Exclusion Criteria:

* Age < 18 years old or ≥ 60 years old;
* Previous solid organ or bone marrow transplantation;
* Autoimmune diseases (rheumatoid arthritis, systemic lupus erythematosus, etc.), or hematologic malignancies (leukemia and lymphoma, etc.);
* Received radiotherapy or chemotherapy within the past 30 days, or received immunosuppressant drugs (tripterygium wilfordii, mycophenolate mofetil, cyclophosphamide, FK506, etc.), or continuous treatment with prednisolone more than 10 mg/day (or equivalent doses of the other hormones);
* Unstable angina pectoris or myocardial infarction in the past six months;
* Acute brain injury (traumatic brain injury, subarachnoid hemorrhage, acute ischemic stroke, acute intracranial hemorrhage, acute intracranial infection, etc.);
* Poorly controlled hypertension and congestive heart failure;
* Increased intraocular or intracranial pressure;
* Chronic kidney disease, received continuous renal replacement therapy in the past 30 days, or acute renal failure requiring CRRT;
* Severe chronic liver disease (Child-Pugh class B or C);
* Alcohol dependence, mental illness or severe cognitive impairment;
* Pregnancy or lactation;
* Informed consent is not obtained.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Serum concentration of inflammatory cytokines (0 h) | 0 hour after study inclusion
  Interleukin (IL)-6, tumor necrosis factor (TNF)-α, IL-2, IL-4, IL-10, IL-17A, and interferon (IFN)-γ
Serum concentration of inflammatory cytokines (48 h) | 48 hours after study inclusion
  IL-6, TNF-α, IL-2, IL-4, IL-10, IL-17A, and IFN-γ
Serum concentration of inflammatory cytokines (72 h) | 72 hours after study inclusion
  IL-6, TNF-α, IL-2, IL-4, IL-10, IL-17A, and IFN-γ
Absolute number of lymphocyte subsets in the peripheral blood (0 h) | 0 hour after study inclusion
  CD3(+), CD3(+) CD4(+), CD3(+) CD8(+), CD3(-) CD16(+) CD56(+) , and CD19(+) cells
Absolute number of lymphocyte subsets in the peripheral blood (48 h) | 48 hours after study inclusion
  CD3(+), CD3(+) CD4(+), CD3(+) CD8(+), CD3(-) CD16(+) CD56(+) , and CD19(+) cells
Absolute number of lymphocyte subsets in the peripheral blood (72 h) | 72 hours after study inclusion
  CD3(+), CD3(+) CD4(+), CD3(+) CD8(+), CD3(-) CD16(+) CD56(+) , and CD19(+) cells
ICU length of stay | up to 8 weeks
  Length of stay in the ICU

SECONDARY OUTCOMES:
Serum concentration of atrial natriuretic peptide (ANP) (0 h) | 0 hour after study inclusion
  ANP is secreted primarily by atrial cardiomyocytes
Serum concentration of atrial natriuretic peptide (ANP) (48h) | 48 hours after study inclusion
  ANP is secreted primarily by atrial cardiomyocytes
Serum concentration of atrial natriuretic peptide (ANP) (72h) | 72 hours after study inclusion
  ANP is secreted primarily by atrial cardiomyocytes
Acute physiology and chronic health evaluation (APACHE) Ⅱ score | 0 hour after study inclusion
  0-67, higher scores correspond to more severe disease and a higher risk of death
Acute physiology and chronic health evaluation (APACHE) Ⅱ score | 24 hours after study inclusion
  0-67, higher scores correspond to more severe disease and a higher risk of death
Acute physiology and chronic health evaluation (APACHE) Ⅱ score | 48 hours after study inclusion
  0-67, higher scores correspond to more severe disease and a higher risk of death
Acute physiology and chronic health evaluation (APACHE) Ⅱ score | 72 hours after study inclusion
  0-67, higher scores correspond to more severe disease and a higher risk of death
Sequential organ failure assessment (SOFA) score | 0 hour after study inclusion
  0-43, higher scores correspond to more severe sepsis
Sequential organ failure assessment (SOFA) score | 24 hours after study inclusion
  0-43, higher scores correspond to more severe sepsis
Sequential organ failure assessment (SOFA) score | 48 hours after study inclusion
  0-43, higher scores correspond to more severe sepsis
Sequential organ failure assessment (SOFA) score | 72 hours after study inclusion
  0-43, higher scores correspond to more severe sepsis
Mechanical ventilation time after inclusion | Up to 8 weeks
  Patients requiring mechanical ventilation after study inclusion
Total hospital length of stay | Through study completion, an average of 2 year
  Total length of hospital stay
Infection complications | Through study completion, an average of 2 year
  Pulmonary infection, urinary tract infection, bloodstream infections, etc
In-hospital mortality | Through study completion, an average of 2 year
  Mortality rates for the entire period of hospitalization
90-day readmission rate | Through study completion, an average of 2 year
  Percentage of readmission to hospital within 90 days of study inclusion
CCL1 expression in alveolar macrophages (0 h) | 0 hour after study inclusion
  CCL1 expression in alveolar macrophages collected from bronchoalveolar lavage fluid
CCL1 expression in alveolar macrophages (24 h) | 24 hours after study inclusion
  CCL1 expression in alveolar macrophages collected from bronchoalveolar lavage fluid
CCL1 expression in alveolar macrophages (72 h) | 72 hours after study inclusion
  CCL1 expression in alveolar macrophages collected from bronchoalveolar lavage fluid
expression of WNT pathway proteins in alveolar macrophages (0 h) | 0 hour after study inclusion
  Wnt5a, FZD5, b-catenin, Lef1 expression in alveolar macrophages collected from bronchoalveolar lavage fluid
expression of WNT pathway proteins in alveolar macrophages (24 h) | 24 hours after study inclusion
  Wnt5a, FZD5, b-catenin, Lef1 expression in alveolar macrophages collected from bronchoalveolar lavage fluid
expression of WNT pathway proteins in alveolar macrophages (72 h) | 72 hours after study inclusion
  Wnt5a, FZD5, b-catenin, Lef1 expression in alveolar macrophages collected from bronchoalveolar lavage fluid

CONTACTS AND LOCATIONS:
Overall Officials: Shiying Yuan, PhD, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
After the completion of the study, the original data will be sent to the email address: zhjcheng1@163.com, and the password will be provided after the paper is published.
Supporting Information: CSR
Time Frame: Six months after the paper was published
Access Criteria: The raw data supporting the conclusions of this manuscript will be made available by the authors, without undue reservation, to any qualified researcher.